CLINICAL TRIAL: NCT04402333
Title: MIRRORS: Minimally Invasive Robotic Surgery, Role in Optimal Debulking Ovarian Cancer, Recovery & Survival
Brief Title: Minimally Invasive Robotic Surgery, Role in Optimal Debulking Ovarian Cancer, Recovery & Survival
Acronym: MIRRORS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Royal Surrey County Hospital NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: MIRRORS
Record Dates: First submitted 2020-05-11; First posted 2020-05-26 (Actual); Last update posted 2020-09-02 (Actual); Status verified 2020-08

CONDITIONS: Ovarian Cancer; Ovarian Neoplasm; Ovarian Neoplasm Epithelial; Fallopian Tube Cancer; Peritoneal Cancer
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Tumour tissue samples from patients undergoing robotic interval debulking surgery and open interval debulking surgery. Analysis will involve primarily immunohistochemistry but may include extracting Ribonucleic acid (RNA).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Robotic interval debulking surgery: Surgery will commence with an initial assessment with a camera inserted though the belly button. This visual assessment will be used to determine whether it is feasible to proceed with surgery robotically or whether full debulking surgery to zero macroscopic residual disease would be best carried out through an open surgical approach. If an open surgical approach is considered the optimum treatment for the patient and they have consented for this, then this will be done. If there is disease that cannot be removed Robotically after starting by this route, but can be removed via an open incision the surgery will be converted to an open procedure if it is safe to do so. If there are any complications, we may also need to convert to open surgery. The aim of the surgery whether by robotic or open is to remove all visible disease safely.
  Interventions: Procedure: Robotic Interval Debulking Surgery
- Open interval debulking surgery: Standard Care. Following initial laparoscopic assessment patients not deemed suitable for minimally invasive robotic surgery will proceed with standard open interval debulking surgery through an extended midline incision. These patients will also be followed up to assess recovery, complication rate and quality of life.

INTERVENTIONS:
Procedure: Robotic Interval Debulking Surgery — Interval debulking surgery carried out in a minimally invasive manner using the Da Vinci Robot.
  Groups: Robotic interval debulking surgery

SUMMARY:
MIRRORS "Minimally Invasive Robotic Surgery, Role in Optimal Debulking Ovarian Cancer, Recovery & Survival" is a new United Kingdom based prospective feasibility study the purpose of which is to establish the feasibility of launching a British multicentre randomised control trial of Robotic interval debulking surgery for ovarian cancer (including cancer of the fallopian tube & peritoneum) in the future. This initial feasibility study will focus on the ability to recruit patients, acceptability, quality of life, the rate at which it is possible to remove all visible tumour and the rate of conversion to open surgery. Ultimately the investigators would like to determine whether, in selected patients, robotic surgery offers improved quality of life and recovery with equivalent overall and progression free survival.

Robotic surgery is unlikely to be suitable in all cases of ovarian cancer, particularly those with large pelvic masses or extensive disease around the upper part of the abdomen, however, it has the potential to provide significant recovery and quality of life benefits to a selected group of patients.

MIRRORS - ICG "Peritoneal angiography / perfusion assessment using Indocyanine green (ICG) in patients with advanced ovarian cancers" is a ancillary study within MIRRORS. Using ICG dye, the investigators aim to observe whether there are any changes in the blood vessel pattern associated with the tumour deposits the investigators remove that makes them distinctive. The ICG will not be used to guide where biopsies are taken or tissue is removed. Participation in this ancillary research is not required for participation in the trial.

DETAILED DESCRIPTION:
Hypothesis: in selected cases of ovarian cancer, following neoadjuvant chemotherapy, minimally invasive robotic surgery provides maximal debulking surgery and improved patient outcomes.

Null Hypothesis: Robotic surgery is not suitable for the treatment of ovarian cancer following neoadjuvant chemotherapy. It is not possible to achieve maximal debulking surgery and patient outcomes are not improved.

To assess the feasibility of obtaining consent from women and acceptability of Robotic interval debulking surgery for advanced ovarian cancer. Women deemed suitable for interval debulking surgery will be identified through the Gynaecological Oncology multidisciplinary team meeting. The aim is to recruit women over a period of 1 year aiming for a total of 20 women who undergo Minimally Invasive Robotic Interval debulking surgery for advanced ovarian cancer. The main outcomes are feasibility of the recruitment process and acceptability of the questionnaires and numeric rating pain scale (NRS11) as assessed by completion rate and patient interviews.

In order to be able to offer MIRRORS to as many patients as possible the investigators have kept the inclusion criteria wide, not restricting by Body Mass Index (BMI), patient comorbidities or Ca125 level.

ELIGIBILITY:
Inclusion Criteria:

Adult women ≥18 years with Stage IIIc -IVb Ovarian cancer (including fallopian tube and peritoneal cancer) undergoing Neo-adjuvant Chemotherapy.

Considered suitable for Interval debulking surgery

≤8cm pelvic mass

MIRRORS ICG Inclusion Criteria - Same as above

Exclusion Criteria:

Pelvic mass >8cm, open surgical approach considered necessary following MDT review. Lacking capacity to the extent they are unable to understand or complete trial documentation / questionnaires.

MIRRORS ICG Exclusion criteria will be:

Severe renal insufficiency estimated Glomerular filtration rate (GFR)< 55ml/min, known allergy to iodine or Indocyanine green (ICG) and hyperthyroidism.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Suitable participants will be identified during the Royal Surrey NHS Foundation Trust Gynaecological Oncology multidisciplinary team meeting (MDT).
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2020-06-26 (Actual); Primary Completion 2021-10-03 (Estimated); Study Completion 2021-10-03 (Estimated)

PRIMARY OUTCOMES:
Recruitment | Assessed at 1 year (recruitment period)
  Number of patients consented compared to the number identified by multidisciplinary team as eligible for inclusion in the study expressed as a percentage.
  Success criteria: At least 20% of people eligible for the study will accept inclusion in the study.

SECONDARY OUTCOMES:
Quality of Life following Surgery | 3 months post surgery
  Assessed using European Organisation for Research and Treatment of Cancer (EORTC) Validated quality of life questionnaire (QLQ) for ovarian cancer (QLQ-C30/QLQ-OV28). This validated questionnaire consists of the core module and its associated ovarian cancer specific module.
Mental wellbeing | 3 months post surgery
  Hospital anxiety and depression scale (HADS) A (Anxiety) and D (Depression) scores are calculated separately. 0-7 = Normal, 8-10 = Borderline, 11-21 = Abnormal (case)
Pain assessment | 3 months post surgery
  Numeric rating scale (NRS11) 0 (no pain) - 10 (worst pain)
Surgical complications | Assessed at close of trial - 15 months +/- 7 days (recruitment + follow up period period) (Quarterly reports to be submitted to sponsor)
  Intraoperative complications will be recorded. Post operative complications will be recorded and classified by Clavien-Dindo Classification.
  Success criteria: Complication rate is not higher than for open interval debulking surgery
Rate of Conversion to open surgery | Assessed at 1 year 3 months (once last recruited patient has undergone surgery)
  Percentage of patients converted to open surgery after being deemed suitable for Robotic interval debulking surgery following initial diagnostic laparoscopy.
  Success criteria: Conversion to open surgery rate not greater than 50% in patient group deemed suitable for Robotic interval debulking surgery following initial diagnostic laparoscopy.
Robotic interval debulking - Maximal Macroscopic debulking rate (R=0 rate) | Assessed at 1 year 3 months (once last recruited patient has undergone surgery)
  Percentage of patients undergoing robotic interval debulking surgery who achieve Maximal macroscopic debulking i.e. no macroscopic residual disease present (R=0 rate)
Overall Survival | Assessed at close of trial - 15 months +/- 7 days (recruitment + follow up period period) reassessed at 5 years to maximum of 10 years
  Measured in Months from the date of surgery.
  In order to follow up long-term survival in participants suffering from ovarian cancer and subsequently correlate this to the research findings it is necessary to store minimal personal data after completion of the study this is detailed in documentation submitted and approved by London - Riverside Research Ethics Committee.
Progression free survival | Assessed at close of trial - 15 months +/- 7 days (recruitment + follow up period period) reassessed at 5 years to maximum of 10 years
  Measured in Months from the date of surgery until the date of first documented progression.
  In order to follow up progression free survival in participants suffering from ovarian cancer and subsequently correlate this to the research findings it is necessary to store minimal personal data after completion of the study this is detailed in documentation submitted and approved by London - Riverside Research Ethics Committee.
Cost | Assessed at close of trial - 15 months +/- 7 days (recruitment + follow up period period)
  Cost of Robotic minimally invasive interval debulking surgery to the hospital compared to a similar open procedure measured in British Pound (GBP) £

CONTACTS AND LOCATIONS:
Overall Officials: Simon Butler-Manuel, MD, Principal Investigator — Royal Surrey NHS Foundation Trust
Locations (1):
- Royal Surrey NHS Foundation Trust, Guildford, Surrey, United Kingdom

IPD SHARING:
Plan to Share IPD: No